CLINICAL TRIAL: NCT06913361
Title: Effects of Gongs Mobilization vs Reverse Distraction Technique in Diabetic Patients With Adhesive Capsulitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/791
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gongs Mobilization (Experimental)
  Interventions: Diagnostic Test: Gongs Mobilization
- Reverse Distraction Technique (Experimental)
  Interventions: Combination Product: Reverse Distraction Technique

INTERVENTIONS:
Diagnostic Test: Gongs Mobilization — The treatment begins with moist heat for 10 minutes, Gong's mobilization with conventional therapy for 8 minutes. The total treatment time was 45 minutes once a day for four days per week for four weeks.
  Arms: Gongs Mobilization
Combination Product: Reverse Distraction Technique — The treatment begins with moist heat for 10 minutes, Reverse Distraction technique with conventional therapy for 8 minutes. The total treatment time was 45 minutes once a day for four days per week for four weeks. Position of the patient: side-lying. The patient is lying at the plinth's edge on the unaffected side. In front of the patient is the therapist's position.
  Arms: Reverse Distraction Technique

SUMMARY:
Adhesive capsulitis (AC) represents a renowned musculoskeletal condition which has been clinically classified as frozen shoulder (FS). Adhesive capsulitis occurs 3-5% of the time in the general population, but in diabetics, the frequency can reach 20%. This study is being conducted to determine the effects of gongs mobilization vs reverse distraction technique in diabetic patients with adhesive capsulitis. This study will be a randomized control trial and data will be collected from Haq Orthopedic Hospital. Sample size is 20 calculated by using G power and adding 20 % attrition.

DETAILED DESCRIPTION:
Non-Probability convenient sampling will be used. Participants meeting the inclusion and exclusion criteria will be divided into two groups.10 subjects in group A will be treated Gongs mobilization and group B will be treated with Reverse distraction technique. Conventional therapy will be given to both groups as base line treatment. Both groups have 4 sessions per week for 4 weeks. All participants will be evaluated before and after the treatment using Numeric Pain Rating scale (NPRS), Shoulder pain and Disability Index (SPADI) and goniometer.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females.
* Diagnosed case of Unilateral Adhesive Capsulitis.
* Age group of 40-60 years.
* Stage 2 and 3 of Adhesive Capsulitis.
* Diabetes Mellitus Type II.
* Patients with decreased ROM (less than or equal to 120 degrees), pain, and mild to moderate levels of type II diabetics (below or equal to 200 mg/dL).
* No history of shoulder surgeries to the affected shoulder.

Exclusion Criteria:

* Systemic arthritic conditions of the shoulder (Rheumatoid arthritis, osteoporosis or malignancies in the shoulder region) .
* Disorders of the Cervical spine .
* Corticosteroids injections in the affected Shoulder in preceding 6 weeks.
* Skin lesions or bruises around the Shoulder.
* Shoulder injuries such as Rotator cuff tear.
* Fracture in and around the shoulder joint.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
NUMERIC PAIN RATING SCALE (NPRS) | 12 Months
  Value of sensitivity/specificity/ validity/reliability: intra-class correlation coefficient 0.58 to 0.93. Measurement: Numerical Interpretation: The Numeric Pain Rating Scale (NPRS) is a simple and widely used tool for assessing pain intensity. Patients rate their pain on a scale from 0 to 10, where 0 indicates ""no pain"" and 10 indicates ""worst pain imaginable."" The interpretation of NPRS scores helps classify pain severity and monitor changes over time.
SHOULDER PAIN AND DISABILITY INDEX | 12 Months
  The items of the questionnaire are assessed on a 0-10 numeric rating scale in which 0 means no disability and 10 is maximum disability. The sum of the seven items equals the total score of the PDI, which ranges from 0 to 70, with higher scores reflecting higher interference of pain with daily activities

CONTACTS AND LOCATIONS:
Locations (1):
- Haq Orthopaedic hospital, Sanda road, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No